CLINICAL TRIAL: NCT00209547
Title: A Phase III, Randomized, Open-Label Study to Assess the Safety and Efficacy of AQUAVAN® Injection Versus Midazolam HCl for Sedation in Patients Undergoing Percutaneous Coronary (PC) Procedures
Brief Title: Study to Assess Safety and Efficacy of AQUAVAN® Injection for Sedation During Cardiac Catheterization
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Collaborators: PPD Development, LP (Industry); Covance (Industry)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 3000-0411
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2008-11-07 (Estimated); Status verified 2008-11

CONDITIONS: Angioplasty; Coronary Catheterization
Keywords: AQUAVAN® Injection; Midazolam; Angioplasty; Coronary catheterization
MeSH Terms: interventions — fospropofol

INTERVENTIONS:
Drug: fospropofol disodium

SUMMARY:
The anticipation of pain and discomfort, a diagnosis, and other intrinsic unknowns make patients anxious both prior to and during a procedure. Therefore, the main goal of sedation with analgesia used during various diagnostic, therapeutic, or surgical procedures is to relieve this anxiety, discomfort, and pain, which are all interrelated. The optimal level of sedation for any given patient is one that allows the patient to tolerate the procedure and provides an appropriate safety margin. This was a study designed to examine the safety and efficacy of AQUAVAN® Injection versus a commonly used approved sedative drug, midazolam HCl following pretreatment with fentanyl citrate injection (for pain relief) in producing sedation in patients undergoing single cardiac catheterization procedures.

DETAILED DESCRIPTION:
This was a randomized, open-label study designed to assess the safety and efficacy of AQUAVAN® Injection (hereafter referred to as AQUAVAN) versus the reference drug, midazolam HCl (hereafter referred to as midazolam) following pretreatment with fentanyl citrate injection (hereafter referred to as fentanyl) in producing sedation in male and female patients undergoing single PC procedures.

Screening assessments were done within 2 weeks of scheduled procedures. After completion of preprocedural sedation assessments, patients were randomly assigned to 1 of the 2 treatment groups at a 3:1 (AQUAVAN: midazolam) allocation ratio on the day of the scheduled procedure (Day 0) via an Interactive Voice Response System (IVRS). Randomization was stratified by site.

All patients, regardless of treatment group assignment, received fentanyl as an analgesic pretreatment. Supplemental doses of fentanyl could be administered if the patient reported pain or if analgesia was inadequate, as demonstrated by increased heart rate and/or blood pressure in the presence of adequate sedation. At no time was fentanyl to be administered to increase sedation levels.

AQUAVAN or midazolam was administered by intravenous (i.v.) bolus to induce a state of minimal-to-moderate (procedural) s sedation, defined as a score of ≤4 on the Modified Observer's Assessment of Alertness/Sedation (OAA/S) scale. Supplemental doses were administered, if necessary, to increase the depth or duration of sedation. Supplemental doses were not administered if the Modified OAA/S score was ≤2 or if there was no purposeful response to stimulation. Patient and Investigator assessments were used to confirm that the depth of sedation met the goals of sedation, reduced anxiety, and awareness.

Follow-up patient assessments were conducted in a telephone interview 24 hours following treatment and during a clinic visit 2 to 5 days following treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patient provided signed/dated Informed Consent and HIPAA authorization after receiving a full explanation of the extent and nature of the study.
2. Patient was at least 18 years of age at the time of screening (Prior to Amendment 2 [dated 04 February 2005], the patient was required to be between 18 and 65 years of age, inclusive. Three subjects were randomized under this earlier inclusion criteria).
3. If female, patient was surgically sterile, postmenopausal or not pregnant or lactating and had been using an acceptable method of birth control for at least 1 month prior to dosing, with a negative urine pregnancy test result at Screening and Predosing Periods.
4. Patient met American Society of Anesthesiologists (ASA)13, 14 Physical Status Classification System level I to III; and
5. Patient was an inpatient or outpatient scheduled to undergo a single PC procedure.

Exclusion Criteria:

1. Patient had history of allergic reaction or hypersensitivity to any anesthetic agent, narcotic, or benzodiazepine.
2. Patient did not meet nils per os (NPO) status per ASA Guideline or institution's guideline.
3. Patient had a condition(s) that, in the opinion of the Investigator, could interfere with appropriate airway management.
4. Patient had participated in an investigational drug study within 1 month prior to study start.
5. Patient had history of mental or visual impairment that would not permit successful measurement of cognitive evaluations.
6. Patient was unwilling to adhere to pre- and postprocedural instructions; or
7. Patient for whom the use of fentanyl or midazolam was contraindicated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110
Dates: Start 2004-02; Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
Demonstrate that AQUAVAN was effective in providing adequate sedation in patients undergoing percutaneous coronary (PC) procedures.

SECONDARY OUTCOMES:
Treatment-emergent adverse events, Sedation-related adverse events, and airway Assistance.

CONTACTS AND LOCATIONS:
Overall Officials: James Jones, MD,PharmD, Study Director — Eisai Inc.